CLINICAL TRIAL: NCT03445273
Title: Maintenance Of aNtiplatElet Therapy in Patients With Coronary Stenting Undergoing Surgery
Acronym: MONET
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Italian Society of Invasive Cardiology (Other)
Responsible Party: Sponsor
Other Study IDs: 11/01/2018
Record Dates: First submitted 2018-02-16; First posted 2018-02-26 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-07

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The MONET registry will include any patient with previous coronary stenting undergoing any type of surgery or operative endoscopic/endovascular procedure. The effects of the application of the Consensus Document "Stent and Surgery-2" on perioperative antiplatelet therapy will be assessed. The study will also assess ischemic and hemorrhagic events in relation to the application of the Consensus Document and length of any antiplatelet discontinuation and delay in performing surgical procedures.

DETAILED DESCRIPTION:
The MONET registry will include any patient with previous coronary stenting undergoing any type of surgery or operative endoscopic/endovascular procedure at the participating Centers. Centers will be divided into two groups: Centers that routinely follow the recommendations of the SAS 2 Document and Centers that do not. The relevant clinical, procedural and outcome data (within index admission and at 30 days) will be entered in a specifically designed electronic case record form (eCRF). The primary endpoint will be the rate of discontinuation of P2Y12 inhibitors and/or aspirin (without bridging) in the first 3 months after PCI with low risk characteristics and 6 months after PCI with high risk characteristics or any antiplatelet therapy discontinuation without bridging therapy. The secondary end-point will be the composite of death, myocardial infarction, probable/definite stent thrombosis and bleeding events at 30 days; the type and the length of discontinuation of any antiplatelet therapy in patients undergoing surgery according to time from PCI to surgery; delay in performing surgical procedure; rate of surgical procedures within 12 months from PCI divided into quartiles (0-3, 3-6, 6-9, 9-12 months).

ELIGIBILITY:
Inclusion Criteria:

* Eligible will be male and female patients > 18 years of age.
* Eligible will be patients with previous coronary stenting undergoing any kind of surgical or operative endoscopic procedure at the participating Centers, irrespective of the distance in time between stenting and surgery.
* Both candidates to elective and urgent/emergent surgical procedures will be included in the MONET registry.

Exclusion Criteria:

* Unwillingness/inability to sign the Informed Consent Form (ICF). Patients with an active bleeding requiring discontinuation of one or both antiplatelet agents will be also excluded. There are no other exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with prior percutaneous coronary intervention (PCI) with stent implantation undergoing urgent or elective surgical/endoscopic procedures
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2018-11-21 (Estimated); Primary Completion 2019-02-21 (Estimated); Study Completion 2019-11-20 (Estimated)

PRIMARY OUTCOMES:
Antiplatelet therapy discontinuation in patients with coronary stenting undergoing surgery | 3 months
  Rate of discontinuation of P2Y12 inhibitors and/or aspirin (without bridging) in the first 3 months after PCI with low risk characteristics and 6 months after PCI with high risk characteristics or any antiplatelet therapy discontinuation without bridging therapy
Antiplatelet therapy discontinuation in patients with coronary stenting undergoing surgery | 6 months
  Rate of discontinuation of P2Y12 inhibitors and/or aspirin (without bridging) in the first 6 months after PCI with high risk characteristics or any antiplatelet therapy discontinuation without bridging therapy

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Musumeci, MD, Principal Investigator — A.O. Santa Croce e Carle di Cuneo, 26 - 12100 - Cuneo (CN)
Locations (5):
- Italy (5):
  - A.O. Santa Croce e Carle di Cuneo, Cuneo, CN
  - Istituto Clinico Humanitas, Rozzano, MI
  - Ospedale degli Infermi, Rivoli, TO
  - A.O. di Cosenza, Cosenza
  - Università Campus Bio-Medico di Roma, Roma

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make Individual Participant Data available

REFERENCES:
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Soliman EZ, Sorlie PD, Sotoodehnia N, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2012 update: a report from the American Heart Association. Circulation. 2012 Jan 3;125(1):e2-e220. doi: 10.1161/CIR.0b013e31823ac046. Epub 2011 Dec 15. No abstract available. PMID 22179539
- [Background] Moschovitis A, Cook S, Meier B. Percutaneous coronary interventions in Europe in 2006. EuroIntervention. 2010 Jun;6(2):189-94. doi: 10.4244/EIJV7I6A31. PMID 20562067
- [Background] Savonitto S, Caracciolo M, Cattaneo M, DE Servi S. Management of patients with recently implanted coronary stents on dual antiplatelet therapy who need to undergo major surgery. J Thromb Haemost. 2011 Nov;9(11):2133-42. doi: 10.1111/j.1538-7836.2011.04456.x. PMID 21819537
- [Background] Authors/Task Force members; Windecker S, Kolh P, Alfonso F, Collet JP, Cremer J, Falk V, Filippatos G, Hamm C, Head SJ, Juni P, Kappetein AP, Kastrati A, Knuuti J, Landmesser U, Laufer G, Neumann FJ, Richter DJ, Schauerte P, Sousa Uva M, Stefanini GG, Taggart DP, Torracca L, Valgimigli M, Wijns W, Witkowski A. 2014 ESC/EACTS Guidelines on myocardial revascularization: The Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS)Developed with the special contribution of the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eur Heart J. 2014 Oct 1;35(37):2541-619. doi: 10.1093/eurheartj/ehu278. Epub 2014 Aug 29. No abstract available. PMID 25173339
- [Background] Patel MR, Dehmer GJ, Hirshfeld JW, Smith PK, Spertus JA; American College of Cardiology Foundation Appropriateness Criteria Task Force; Society for Cardiovascular Angiography and Interventions; Society of Thoracic Surgeons; American Association for Thoracic Surgery; American Heart Association, and the American Society of Nuclear Cardiology Endorsed by the American Society of Echocardiography; Heart Failure Society of America; Society of Cardiovascular Computed Tomography. ACCF/SCAI/STS/AATS/AHA/ASNC 2009 Appropriateness Criteria for Coronary Revascularization: a report by the American College of Cardiology Foundation Appropriateness Criteria Task Force, Society for Cardiovascular Angiography and Interventions, Society of Thoracic Surgeons, American Association for Thoracic Surgery, American Heart Association, and the American Society of Nuclear Cardiology Endorsed by the American Society of Echocardiography, the Heart Failure Society of America, and the Society of Cardiovascular Computed Tomography. J Am Coll Cardiol. 2009 Feb 10;53(6):530-53. doi: 10.1016/j.jacc.2008.10.005. PMID 19195618
- [Background] McFadden EP, Stabile E, Regar E, Cheneau E, Ong AT, Kinnaird T, Suddath WO, Weissman NJ, Torguson R, Kent KM, Pichard AD, Satler LF, Waksman R, Serruys PW. Late thrombosis in drug-eluting coronary stents after discontinuation of antiplatelet therapy. Lancet. 2004 Oct 23-29;364(9444):1519-21. doi: 10.1016/S0140-6736(04)17275-9. PMID 15500897
- [Background] Iakovou I, Schmidt T, Bonizzoni E, Ge L, Sangiorgi GM, Stankovic G, Airoldi F, Chieffo A, Montorfano M, Carlino M, Michev I, Corvaja N, Briguori C, Gerckens U, Grube E, Colombo A. Incidence, predictors, and outcome of thrombosis after successful implantation of drug-eluting stents. JAMA. 2005 May 4;293(17):2126-30. doi: 10.1001/jama.293.17.2126. PMID 15870416
- [Background] Spertus JA, Kettelkamp R, Vance C, Decker C, Jones PG, Rumsfeld JS, Messenger JC, Khanal S, Peterson ED, Bach RG, Krumholz HM, Cohen DJ. Prevalence, predictors, and outcomes of premature discontinuation of thienopyridine therapy after drug-eluting stent placement: results from the PREMIER registry. Circulation. 2006 Jun 20;113(24):2803-9. doi: 10.1161/CIRCULATIONAHA.106.618066. Epub 2006 Jun 12. PMID 16769908
- [Background] van Werkum JW, Heestermans AA, Zomer AC, Kelder JC, Suttorp MJ, Rensing BJ, Koolen JJ, Brueren BR, Dambrink JH, Hautvast RW, Verheugt FW, ten Berg JM. Predictors of coronary stent thrombosis: the Dutch Stent Thrombosis Registry. J Am Coll Cardiol. 2009 Apr 21;53(16):1399-409. doi: 10.1016/j.jacc.2008.12.055. PMID 19371823
- [Background] Park DW, Park SW, Park KH, Lee BK, Kim YH, Lee CW, Hong MK, Kim JJ, Park SJ. Frequency of and risk factors for stent thrombosis after drug-eluting stent implantation during long-term follow-up. Am J Cardiol. 2006 Aug 1;98(3):352-6. doi: 10.1016/j.amjcard.2006.02.039. Epub 2006 Jun 12. PMID 16860022
- [Background] Kaluza GL, Joseph J, Lee JR, Raizner ME, Raizner AE. Catastrophic outcomes of noncardiac surgery soon after coronary stenting. J Am Coll Cardiol. 2000 Apr;35(5):1288-94. doi: 10.1016/s0735-1097(00)00521-0. PMID 10758971
- [Background] Akowuah E, Shrivastava V, Jamnadas B, Hopkinson D, Sarkar P, Storey R, Braidley P, Cooper G. Comparison of two strategies for the management of antiplatelet therapy during urgent surgery. Ann Thorac Surg. 2005 Jul;80(1):149-52. doi: 10.1016/j.athoracsur.2005.01.009. PMID 15975358
- [Background] Rossini R, Capodanno D, Lettieri C, Musumeci G, Nijaradze T, Romano M, Lortkipanidze N, Cicorella N, Biondi Zoccai G, Sirbu V, Izzo A, Guagliumi G, Valsecchi O, Gavazzi A, Angiolillo DJ. Prevalence, predictors, and long-term prognosis of premature discontinuation of oral antiplatelet therapy after drug eluting stent implantation. Am J Cardiol. 2011 Jan 15;107(2):186-94. doi: 10.1016/j.amjcard.2010.08.067. PMID 21211596
- [Background] To AC, Armstrong G, Zeng I, Webster MW. Noncardiac surgery and bleeding after percutaneous coronary intervention. Circ Cardiovasc Interv. 2009 Jun;2(3):213-21. doi: 10.1161/CIRCINTERVENTIONS.108.830158. Epub 2009 Apr 21. PMID 20031718
- [Background] Cutlip DE, Baim DS, Ho KK, Popma JJ, Lansky AJ, Cohen DJ, Carrozza JP Jr, Chauhan MS, Rodriguez O, Kuntz RE. Stent thrombosis in the modern era: a pooled analysis of multicenter coronary stent clinical trials. Circulation. 2001 Apr 17;103(15):1967-71. doi: 10.1161/01.cir.103.15.1967. PMID 11306525
- [Background] Patrono C, Bachmann F, Baigent C, Bode C, De Caterina R, Charbonnier B, Fitzgerald D, Hirsh J, Husted S, Kvasnicka J, Montalescot G, Garcia Rodriguez LA, Verheugt F, Vermylen J, Wallentin L, Priori SG, Alonso Garcia MA, Blanc JJ, Budaj A, Cowie M, Dean V, Deckers J, Fernandez Burgos E, Lekakis J, Lindahl B, Mazzotta G, Morais J, Oto A, Smiseth OA, Morais J, Deckers J, Ferreira R, Mazzotta G, Steg PG, Teixeira F, Wilcox R; European Society of Cardiology. Expert consensus document on the use of antiplatelet agents. The task force on the use of antiplatelet agents in patients with atherosclerotic cardiovascular disease of the European society of cardiology. Eur Heart J. 2004 Jan;25(2):166-81. doi: 10.1016/j.ehj.2003.10.013. No abstract available. PMID 14720534
- [Background] Abualsaud AO, Eisenberg MJ. Perioperative management of patients with drug-eluting stents. JACC Cardiovasc Interv. 2010 Feb;3(2):131-42. doi: 10.1016/j.jcin.2009.11.017. PMID 20170869
- [Background] Kumar R, McKinney WP, Raj G, Heudebert GR, Heller HJ, Koetting M, McIntire DD. Adverse cardiac events after surgery: assessing risk in a veteran population. J Gen Intern Med. 2001 Aug;16(8):507-18. doi: 10.1046/j.1525-1497.2001.016008507.x. PMID 11556926
- [Background] Badner NH, Knill RL, Brown JE, Novick TV, Gelb AW. Myocardial infarction after noncardiac surgery. Anesthesiology. 1998 Mar;88(3):572-8. doi: 10.1097/00000542-199803000-00005. PMID 9523798
- [Background] Shah KB, Kleinman BS, Rao TL, Jacobs HK, Mestan K, Schaafsma M. Angina and other risk factors in patients with cardiac diseases undergoing noncardiac operations. Anesth Analg. 1990 Mar;70(3):240-7. doi: 10.1213/00000539-199003000-00002. PMID 2305974
- [Background] Srinivasan AK, Grayson AD, Pullan DM, Fabri BM, Dihmis WC. Effect of preoperative aspirin use in off-pump coronary artery bypass operations. Ann Thorac Surg. 2003 Jul;76(1):41-5. doi: 10.1016/s0003-4975(03)00182-6. PMID 12842510
- [Background] Ferraris VA, Ferraris SP, Moliterno DJ, Camp P, Walenga JM, Messmore HL, Jeske WP, Edwards FH, Royston D, Shahian DM, Peterson E, Bridges CR, Despotis G; Society of Thoracic Surgeons. The Society of Thoracic Surgeons practice guideline series: aspirin and other antiplatelet agents during operative coronary revascularization (executive summary). Ann Thorac Surg. 2005 Apr;79(4):1454-61. doi: 10.1016/j.athoracsur.2005.01.008. No abstract available. PMID 15797109
- [Background] Purkayastha S, Athanasiou T, Malinovski V, Tekkis P, Foale R, Casula R, Glenville B, Darzi A. Does clopidogrel affect outcome after coronary artery bypass grafting? A meta-analysis. Heart. 2006 Apr;92(4):531-2. doi: 10.1136/hrt.2004.058396. No abstract available. PMID 16537769
- [Background] Ascione R, Ghosh A, Rogers CA, Cohen A, Monk C, Angelini GD. In-hospital patients exposed to clopidogrel before coronary artery bypass graft surgery: a word of caution. Ann Thorac Surg. 2005 Apr;79(4):1210-6. doi: 10.1016/j.athoracsur.2004.09.046. PMID 15797051
- [Background] Yende S, Wunderink RG. Effect of clopidogrel on bleeding after coronary artery bypass surgery. Crit Care Med. 2001 Dec;29(12):2271-5. doi: 10.1097/00003246-200112000-00006. PMID 11801823
- [Background] Chu MW, Wilson SR, Novick RJ, Stitt LW, Quantz MA. Does clopidogrel increase blood loss following coronary artery bypass surgery? Ann Thorac Surg. 2004 Nov;78(5):1536-41. doi: 10.1016/j.athoracsur.2004.03.028. PMID 15511426
- [Background] Leong JY, Baker RA, Shah PJ, Cherian VK, Knight JL. Clopidogrel and bleeding after coronary artery bypass graft surgery. Ann Thorac Surg. 2005 Sep;80(3):928-33. doi: 10.1016/j.athoracsur.2005.03.074. PMID 16122457
- [Background] Burger W, Chemnitius JM, Kneissl GD, Rucker G. Low-dose aspirin for secondary cardiovascular prevention - cardiovascular risks after its perioperative withdrawal versus bleeding risks with its continuation - review and meta-analysis. J Intern Med. 2005 May;257(5):399-414. doi: 10.1111/j.1365-2796.2005.01477.x. PMID 15836656
- [Background] Gurbel PA, DiChiara J, Tantry US. Antiplatelet therapy after implantation of drug-eluting stents: duration, resistance, alternatives, and management of surgical patients. Am J Cardiol. 2007 Oct 22;100(8B):18M-25M. doi: 10.1016/j.amjcard.2007.08.018. PMID 17950828
- [Background] Chassot PG, Delabays A, Spahn DR. Perioperative antiplatelet therapy: the case for continuing therapy in patients at risk of myocardial infarction. Br J Anaesth. 2007 Sep;99(3):316-28. doi: 10.1093/bja/aem209. Epub 2007 Jul 23. PMID 17650517
- [Background] Brilakis ES, Banerjee S, Berger PB. Perioperative management of patients with coronary stents. J Am Coll Cardiol. 2007 Jun 5;49(22):2145-50. doi: 10.1016/j.jacc.2007.02.046. Epub 2007 May 23. PMID 17543633
- [Background] Riddell JW, Chiche L, Plaud B, Hamon M. Coronary stents and noncardiac surgery. Circulation. 2007 Oct 16;116(16):e378-82. doi: 10.1161/CIRCULATIONAHA.107.726992. No abstract available. PMID 17938292
- [Background] Fleisher LA, Beckman JA, Brown KA, Calkins H, Chaikof EL, Fleischmann KE, Freeman WK, Froehlich JB, Kasper EK, Kersten JR, Riegel B, Robb JF, Smith SC Jr, Jacobs AK, Adams CD, Anderson JL, Antman EM, Buller CE, Creager MA, Ettinger SM, Faxon DP, Fuster V, Halperin JL, Hiratzka LF, Hunt SA, Lytle BW, Nishimura R, Ornato JP, Page RL, Riegel B, Tarkington LG, Yancy CW; American College of Cardiology; American Heart Association Task Force on Practice Guidelines (writing Committee to Revise the 2002 Guidelines on Perioperative Cardiovascular Evaluation for Noncardiac Surgery); American Society of Echocardiography; American Society of Nuclear Cardiology; Heart Rhythm Society; Society of Cardiovascular Anesthesiologists; Society for Cardiovascular Angiography and Interventions; Society for Vascular Medicine and Biology; Society for Vascular Surgery. ACC/AHA 2007 guidelines on perioperative cardiovascular evaluation and care for noncardiac surgery: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the 2002 Guidelines on Perioperative Cardiovascular Evaluation for Noncardiac Surgery) developed in collaboration with the American Society of Echocardiography, American Society of Nuclear Cardiology, Heart Rhythm Society, Society of Cardiovascular Anesthesiologists, Society for Cardiovascular Angiography and Interventions, Society for Vascular Medicine and Biology, and Society for Vascular Surgery. J Am Coll Cardiol. 2007 Oct 23;50(17):e159-241. doi: 10.1016/j.jacc.2007.09.003. No abstract available. PMID 17950140
- [Background] Eagle KA, Guyton RA, Davidoff R, Edwards FH, Ewy GA, Gardner TJ, Hart JC, Herrmann HC, Hillis LD, Hutter AM Jr, Lytle BW, Marlow RA, Nugent WC, Orszulak TA, Antman EM, Smith SC Jr, Alpert JS, Anderson JL, Faxon DP, Fuster V, Gibbons RJ, Gregoratos G, Halperin JL, Hiratzka LF, Hunt SA, Jacobs AK, Ornato JP; American College of Cardiology; American Heart Association Task Force on Practice Guidelines; American Society for Thoracic Surgery and the Society of Thoracic Surgeons. ACC/AHA 2004 guideline update for coronary artery bypass graft surgery: summary article: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee to Update the 1999 Guidelines for Coronary Artery Bypass Graft Surgery). Circulation. 2004 Aug 31;110(9):1168-76. doi: 10.1161/01.CIR.0000138790.14877.7D. No abstract available. PMID 15339866
- [Background] Grines CL, Bonow RO, Casey DE Jr, Gardner TJ, Lockhart PB, Moliterno DJ, O'Gara P, Whitlow P; American Heart Association; American College of Cardiology; Society for Cardiovascular Angiography and Interventions; American College of Surgeons; American Dental Association; American College of Physicians. Prevention of premature discontinuation of dual antiplatelet therapy in patients with coronary artery stents: a science advisory from the American Heart Association, American College of Cardiology, Society for Cardiovascular Angiography and Interventions, American College of Surgeons, and American Dental Association, with representation from the American College of Physicians. J Am Coll Cardiol. 2007 Feb 13;49(6):734-9. doi: 10.1016/j.jacc.2007.01.003. PMID 17291948
- [Background] Task Force for Preoperative Cardiac Risk Assessment and Perioperative Cardiac Management in Non-cardiac Surgery; European Society of Cardiology (ESC); Poldermans D, Bax JJ, Boersma E, De Hert S, Eeckhout E, Fowkes G, Gorenek B, Hennerici MG, Iung B, Kelm M, Kjeldsen KP, Kristensen SD, Lopez-Sendon J, Pelosi P, Philippe F, Pierard L, Ponikowski P, Schmid JP, Sellevold OF, Sicari R, Van den Berghe G, Vermassen F. Guidelines for pre-operative cardiac risk assessment and perioperative cardiac management in non-cardiac surgery. Eur Heart J. 2009 Nov;30(22):2769-812. doi: 10.1093/eurheartj/ehp337. Epub 2009 Aug 27. No abstract available. PMID 19713421
- [Background] Cardiac Society of Australia and New Zealand. Guidelines for the management of antiplatelet therapy in patients with coronary stents undergoing non-cardiac surgery. Heart Lung Circ. 2010 Jan;19(1):2-10. doi: 10.1016/j.hlc.2009.10.008. Epub 2009 Dec 31. No abstract available. PMID 20045378
- [Background] Samama CM, Bastien O, Forestier F, Denninger MH, Isetta C, Juliard JM, Lasne D, Leys D, Mismetti P; French Society of Anesthesiology and Intensive Care. Antiplatelet agents in the perioperative period: expert recommendations of the French Society of Anesthesiology and Intensive Care (SFAR) 2001--summary statement. Can J Anaesth. 2002 Jun-Jul;49(6):S26-35. PMID 12557412
- [Background] Douketis JD, Spyropoulos AC, Spencer FA, Mayr M, Jaffer AK, Eckman MH, Dunn AS, Kunz R. Perioperative management of antithrombotic therapy: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e326S-e350S. doi: 10.1378/chest.11-2298. PMID 22315266
- [Background] Rossini R, Bramucci E, Castiglioni B, De Servi S, Lettieri C, Lettino M, Musumeci G, Visconti LO, Piccaluga E, Savonitto S, Trabattoni D, Buffoli F, Angiolillo DJ, Bovenzi F, Cremonesi A, Scherillo M, Guagliumi G; Societa Italiana di Cardiologia Invasiva (GISE); Associazione Nazionale Medici Cardiologi Ospedalieri (ANMCO). [Coronary stenting and surgery: perioperative management of antiplatelet therapy in patients undergoing surgery after coronary stent implantation]. G Ital Cardiol (Rome). 2012 Jul-Aug;13(7-8):528-51. doi: 10.1714/1114.12251. Italian. PMID 22781382
- [Background] Cutlip DE, Windecker S, Mehran R, Boam A, Cohen DJ, van Es GA, Steg PG, Morel MA, Mauri L, Vranckx P, McFadden E, Lansky A, Hamon M, Krucoff MW, Serruys PW; Academic Research Consortium. Clinical end points in coronary stent trials: a case for standardized definitions. Circulation. 2007 May 1;115(17):2344-51. doi: 10.1161/CIRCULATIONAHA.106.685313. PMID 17470709
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Writing Group on the Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Thygesen K, Alpert JS, White HD, Jaffe AS, Katus HA, Apple FS, Lindahl B, Morrow DA, Chaitman BA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S; ESC Committee for Practice Guidelines (CPG). Third universal definition of myocardial infarction. Eur Heart J. 2012 Oct;33(20):2551-67. doi: 10.1093/eurheartj/ehs184. Epub 2012 Aug 24. No abstract available. PMID 22922414
- [Background] Devereaux PJ, Xavier D, Pogue J, Guyatt G, Sigamani A, Garutti I, Leslie K, Rao-Melacini P, Chrolavicius S, Yang H, Macdonald C, Avezum A, Lanthier L, Hu W, Yusuf S; POISE (PeriOperative ISchemic Evaluation) Investigators. Characteristics and short-term prognosis of perioperative myocardial infarction in patients undergoing noncardiac surgery: a cohort study. Ann Intern Med. 2011 Apr 19;154(8):523-8. doi: 10.7326/0003-4819-154-8-201104190-00003. PMID 21502650

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-25): https://cdn.clinicaltrials.gov/large-docs/73/NCT03445273/Prot_SAP_000.pdf